CLINICAL TRIAL: NCT07116330
Title: Late-Onset Seizures: Trial of Vascular Risk Investigation and Treatment
Acronym: LOSTIT
Status: Not yet recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Sodra Alvsborgs Hospital (Other); Skane University Hospital (Other); Danderyd Hospital (Other); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Johan Zelano, Professor, Sahlgrenska University Hospital
Other Study IDs: 2024-08662
Record Dates: First submitted 2025-06-10; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy; Seizure
Keywords: vascular risk; cardiovascular
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Blood Pressure; Health Records, Personal; Body Mass Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First seizure after age 50: All patients evaluated for a first seizure after age 50 at the providers.
  Interventions: Other: Vascuar risk factor screening (blood pressure, medical history, BMI, laboratory tests)

INTERVENTIONS:
Other: Vascuar risk factor screening (blood pressure, medical history, BMI, laboratory tests) — The vascular risk assessment is outlined below, there may be slight variations according to local routines. Overall, the screening should include:
  Family history of vascular disease
  Tests/examinations (order or obtain from medical records [past 3 months]) Weight Height Waist circumference 12-lead ECG Resting and standing blood pressure Total cholesterol HDL cholesterol LDL cholesterol HbA1c High sensitivity CRP Serum creatinine Urine albumin-to-creatinine ratio
  Medical history Atherosclerotic cardiovascular disease Atrial fibrillation Congestive heart failure Diabetes mellitus Hypertension Kidney disease Life-style risk factors (smoking, exercis

SUMMARY:
A growing body of evidence suggests patients with late-onset seizures are at an increased risk of stroke, but the potential for reducing cardiovascular morbidity through risk factor screening and management is unknown.

The investigators aim to determine whether individuals with new-onset unprovoked seizures after middle age should undergo vascular risk assessment. In a cluster project the investigators assess the effect of vascular risk factor screening in an observational study as well as a cohort study.

The project has two interlinked components: a prospective single group study, in which risk factor assessment is performed and subsequent management is followed for one year; and a register-based cohort study examining the long-term effects of the intervention on a system level.

DETAILED DESCRIPTION:
Cluster design: Participating sites start with vascular risk factor intervention - patients are then offered participation in an observational 1-year study. In addition, all patients at the sites are followed in registers and compared to historic controls. Follow-up in the register study will be at least 5, but probably 10 years (until significant difference in primary analysis - Kaplan Meier).

ELIGIBILITY:
Inclusion Criteria

Clinical study:

- First assessment for unprovoked seizures or epilepsy with onset after age 50 -- - vascular risk factor evaluation per the new routine at participating care givers

Register study:

* age ≥50 with a first-ever outpatient appointment to one of the participating clinics and
* a first-listed diagnostic code for seizures or epilepsy (ICD-10: R568, G40)

Exclusion Criteria

Clinical study:

* Inability to consent.
* Progressive brain disease (tumour or degenerative)

Register study:

* preexisting seizures/epilepsy, as demonstrated by a registered diagnostic code for seizures (ICD-10: R568, G40, G41) or a dispensed antiseizure medication (ATC-code: N03) more than 3 months before the initial consultation
* a registered diagnostic code for stroke or TIA (ICD-10: I61, I63, I64, or G45 except G454) before the initial consultation, or
* progressive brain disease, as indicated by diagnostic codes or drug prescriptions suggestive of brain tumors (ICD-10: C71, D33, D43, C793) or
* neurocognitive disorders (ICD-10: F00-F03, F051, G30, G318, G912; ATC code: N06D).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥50 with a first-ever outpatient appointment for seizures or epilepsy to one of the participating clinics.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Proportion with pharmacological intervention | 1 year
  The proportion with pharmacological intervention of modifiable vascular risk factors.

SECONDARY OUTCOMES:
Secondary outcomes in prospective clinical study | At recruitment
  Proportion (%) with hypertension, diabetes mellitus, moderate to severe chronic kidney disease, atrial fibrillation.
Secondary outcomes at 1 year follow-up prospective clinical study | 1 year
  Delta (absolute and %) in modifiable vascular risk factors compared to baseline, changes in SCORE2/SCORE2-OP, adverse effects, arrhythmias, retention of pharmacological intervention.

OTHER OUTCOMES:
Register study outcomes | 5-10 years
  The primary outcome is a registered acute stroke, measured with yearly extractions from the Swedish national stroke register (95% coverage of acute strokes in Sweden).
  Secondary outcomes: cardiovascular events, a composite measure of the variables stroke (primary outcome), myocardial infarction (ICD-10 I21-I22 in NPR or death from myocardial infarction in the CDR), and cardiovascular death (an ICD-10 code of I0-I99 [diseases of the circulatory system] as the underlying cause of death). Other secondary outcomes include all-cause mortality, stroke severity (NIHSS at stroke admission; modified Rankin Scale 3 months post-stroke), arrythmias or conduction disorder (relevant ICD-10/procedure codes suggestive of conduction disorder, arrhythmia or cardiac arrest), and occurrence of recurrent seizures, captured by the NPR (hospital admissions [inpatient care] or emergency room visits with a seizure-related diagnostic code [ICD-10: R56.8, G40, or G41] as the first-listed diagnosis).

CONTACTS AND LOCATIONS:
Locations (1):
- Södra Älvsborg Sjukhus, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No
Privacy laws and regulations prevent most sharing of data. Anonymized or processed data may be shared upon reasonable request if regulatory possibilities allow.

REFERENCES:
- [Background] Larsson D, Asberg S, Sundstrom J, Frid P, Zelano J. Cardiovascular risk factor assessment in late-onset seizures: A study protocol to assess the value of structured intervention. Epilepsia Open. 2024 Aug;9(4):1611-1617. doi: 10.1002/epi4.12987. Epub 2024 Jun 14. PMID 38874366